CLINICAL TRIAL: NCT06454513
Title: Exploration on the Efficacy of Different Anesthesia Methods in Transbronchial Biopsy
Brief Title: Efficacy of Different Anesthesia Methods in Transbronchial Biopsy
Acronym: EDAMTBB
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Guanghong Zhou, Department of Respiratory and Critical Care Medicine, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPHGZ03
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia; Respiratory Diseases; Biopsy
Keywords: Anesthesia method; Bronchoscopic biopsy; Efficiency research
MeSH Terms: conditions — Respiratory Tract Diseases | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia: There all cases in this group where the surgical anesthesia method is general anesthesia
  Interventions: Procedure: general anesthesia
- Local anesthesia: There all cases in this group where the surgical anesthesia method is local anesthesia

INTERVENTIONS:
Procedure: general anesthesia — Different anesthesia methods
  Groups: General anesthesia

SUMMARY:
This study investigates the efficacy of different anesthesia methods (general anesthesia with laryngeal mask airway and local nebulized anesthesia) for transbronchial biopsy using an electronic bronchoscope. The study retrospectively analyzed cases of transbronchial biopsy performed at the Respiratory Endoscopy Center of Sichuan Provincial People's Hospital from June 5, 2020, to June 5, 2024. Data collected included age, gender, primary diagnosis, anesthesia method, biopsy method, operation time (excluding general anesthesia and laryngeal mask airway placement time), lesion location and size, pathological results, and follow-up status.

DETAILED DESCRIPTION:
General anesthesia and local anesthesia are the primary anesthesia methods for interventional respiratory endoscopy. While general anesthesia offers greater comfort, it carries anesthesia-related risks. Local anesthesia, on the other hand, provides a relatively low surgical risk and cost-effectiveness. However, there is limited research on whether its diagnostic value is inferior to that of general anesthesia.This study investigates the efficacy of the two anesthesia methods (general anesthesia with laryngeal mask airway and local nebulized anesthesia) for transbronchial biopsy. The study retrospectively analyzed cases of transbronchial biopsy performed at the Respiratory Endoscopy Center of Sichuan Provincial People's Hospital from June 5, 2020, to June 5, 2024. Data collected included age, gender, primary diagnosis, anesthesia method, biopsy method(forcep/cryobiopsy), operation time (excluding general anesthesia and laryngeal mask airway placement time), lesion location and size, pathological results, and follow-up status(pneumothorax、hemorrhage).

ELIGIBILITY:
Inclusion Criteria:

* Completed Transbronchial Biopsy；the platelets count and PT, APTT tests were normal, normal ECG, Anesthesiologist evaluation was needed in General anesthesia group.

Exclusion Criteria:

* patients with contraindication of bronchoscopy (such as respiratory failure and acute cardio-cerebrovascular events), and women who were pregnant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who require biopsy to further clarify the nature of lung lesions
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficacy | baseline
  The diagnostic positivity rate(%) of transbronchial biopsy under different anesthesia methods between two groups

SECONDARY OUTCOMES:
Clinical information | baseline
  age（year）, gender(male/female), primary diagnosis(lung cancer/pneumonia or other)
lesion location (left/right/other) | baseline
  Clinical information
lesion size (mm) | baseline
  Clinical information
Postoperative complications (hemorrhage or pneumothorax） | baseline
  Clinical information
Operation time | intraoperative
  Clinical information

CONTACTS AND LOCATIONS:
Overall Officials: Guanghong G Zhou, Principal Investigator — Sichuan Academy of Medical Sciences
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No